CLINICAL TRIAL: NCT06542835
Title: Community Partnership for Telehealth Solutions to Counter Misinformation and Achieve Equity
Acronym: PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: San Diego State University (Other); AltaMed Health Services Corporation (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Gloria Coronado, Principal Investigator, University of Arizona
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: STUDY00004612
Record Dates: First submitted 2024-07-19; First posted 2024-08-07 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer
Keywords: cancer screening; telehealth; video; text messaging; patient navigation; stool testing; fecal testing; Latinx health disparities
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video text message, mailed FIT, and social needs navigation (Experimental): Tailored video text message, mailed FIT, and navigation to address patients' social needs.
  Interventions: Behavioral: Video text message; Behavioral: Mailed FIT; Behavioral: Social needs navigation
- Usual care (Active Comparator): Colorectal cancer (CRC) screening offers during in-person clinic visits.
  Interventions: Behavioral: In-clinic CRC screening promotion; Behavioral: Reminders

INTERVENTIONS:
Behavioral: Video text message — Video text messages tailored to the Latinx population to educate and motivate patients to complete CRC screening.
  Arms: Video text message, mailed FIT, and social needs navigation
Behavioral: In-clinic CRC screening promotion — Stool-test orders, colonoscopy referrals.
  Arms: Usual care
Behavioral: Mailed FIT — Mailed FIT kits.
  Arms: Video text message, mailed FIT, and social needs navigation
Behavioral: Social needs navigation — Patient navigation to address social needs.
  Arms: Video text message, mailed FIT, and social needs navigation
Behavioral: Reminders — Centralized text and/or telephone reminders for ordered tests.
  Arms: Usual care

SUMMARY:
Non-randomized, two-arm stepped-wedge trial of a multi-level colorectal cancer screening intervention.

DETAILED DESCRIPTION:
The PRIME study aims to improve colorectal cancer (CRC) screening and follow-up among predominantly Latinx populations by using video text messages, mailed FIT kits, and patient navigation. The study will address multi-level barriers to screening, including misinformation, lack of access, and social determinants of health. The hypothesis is that a multi-component intervention will increase CRC screening rates and follow-up care, reducing disparities in CRC outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ages 45-64
* Eligible for colorectal cancer (CRC) screening
* Current patients (seen in the clinic in the last 6 months)
* Primary speaker of English or Spanish
* Cell phone listed in Electronic Health Record (EHR)
* No recent history of CRC screening
* Resides in one of the neighborhoods included in the main trial

Exclusion Criteria:

* Colorectal disease (e.g., ulcerative colitis or colectomy)
* Personal history of colorectal cancer
* End-stage or life-threatening diseases
* Known to be under hospice care
* Living in a skilled nursing facility
* Patients who decline research participation will be removed from the patient contact list

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6000 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
CRC Screening Completion at the Individual Level | 6 months
  Measure the completion rate of colorectal cancer (CRC) screening at the individual level within 6 months of receiving the intervention. This will compare the proportion of participants in the post-intervention group versus the pre-intervention group.

SECONDARY OUTCOMES:
FIT completion | 6 months
  Measure the completion rate of fecal immunochemical tests (FIT) within 6 months of receiving the intervention. This will compare the proportion of participants who complete FIT in the post-intervention group versus the pre-intervention group.
Rate of Follow-Up Colonoscopy Completion | 12 months
  Track the completion rate of follow-up colonoscopy within 12 months for participants with abnormal FIT results, comparing the post-intervention versus pre-intervention groups.
Time to follow-up colonoscopy | Within 12 months post abnormal FIT result
  Measure the time from abnormal FIT result to the completion of follow-up colonoscopy, comparing the post-intervention versus the pre-intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Escaron, PhD, Principal Investigator — AltaMed Health Services Corporation
Locations (1):
- AltaMed Health Services Corporation, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rivelli JS, Schneider JL, Vaughn KA, Locher BW, Shaw MC, Martinez LS, Ruiz E, Thompson JH, Escaron AL, Coronado GD. Improving animated instructional videos for colorectal cancer screening: An application of learner verification and revision. Transl Behav Med. 2025 Jan 16;15(1):ibaf020. doi: 10.1093/tbm/ibaf020. PMID 40526315